CLINICAL TRIAL: NCT02596009
Title: Multicenter Open-label Cross-over Study to Compare Inspiratory Flow Rates Achieved by the COPD Patients Through Breezhaler®, Ellipta® and Handihaler® Dry Powder Inhaler Devices
Brief Title: Inspiratory Flow Rates Achieved by the COPD Patients Through Breezhaler®, Ellipta® and Handihaler® Inhaler Devices
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CNVA237A2403
Record Dates: First submitted 2015-10-14; First posted 2015-11-04 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive (COPD)
Keywords: COPD; Cachexia due to chronic obstructive pulmonary disease; wasting syndrome; Loss of weight; muscle atrophy; loss of body mass; signficant loss of appetite; cachectic syndrome
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive; Wasting Syndrome; Weight Loss; Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Breezhaler® (Experimental): Each patient was required to inhale via Breezhaler® in a randomized cross-over sequence. The randomization numbers were generated using 6 sequences: BEH, EHB, HBE, BHE, EBH, HEB (B: Breezhaler, E: Ellipta, H: Handihaler).
  Interventions: Device: Breezhaler®
- Ellipta® (Other): Each patient were required to inhale via Ellipta® in a randomized cross-over sequence. The randomization numbers were generated using 6 sequences: BEH, EHB, HBE, BHE, EBH, HEB (B: Breezhaler, E: Ellipta, H: Handihaler).
  Interventions: Device: Ellipta®
- Handihaler® (Other): Each patient were required to inhale via Handihaler® in a randomized cross-over sequence. The randomization numbers were generated using 6 sequences: BEH, EHB, HBE, BHE, EBH, HEB (B: Breezhaler, E: Ellipta, H: Handihaler).
  Interventions: Device: Handihaler®

INTERVENTIONS:
Device: Breezhaler® — No active drug or placebo were administered to patients during this study. Each patient were required to inhale via all three (03) study devices (Breezhaler®, Ellipta® and Handihaler®). Each patient was required to produce at least three (03) inhalational profiles via each inhalational device, following the training and demonstration for correct inhalational procedure, for each device.
  Arms: Breezhaler®
Device: Ellipta® — No active drug or placebo were administered to patients during this study. Each patient were required to inhale via all three (03) study devices (Breezhaler®, Ellipta® and Handihaler®). Each patient was required to produce at least three (03) inhalational profiles via each inhalational device, following the training and demonstration for correct inhalational procedure, for each device.
  Arms: Ellipta®
Device: Handihaler® — No active drug or placebo were administered to patients during this study. Each patient were required to inhale via all three (03) study devices (Breezhaler®, Ellipta® and Handihaler®). Each patient was required to produce at least three (03) inhalational profiles via each inhalational device, following the training and demonstration for correct inhalational procedure, for each device.
  Arms: Handihaler®

SUMMARY:
The purpose of this study was to compare dynamic inspiratory flow rates achieved by a population of Chronic Obstructive Pulmonary Disease (COPD) patients through the Breezhaler®, Ellipta® and Handihaler® dry powder inhaler (DPI) devices. No active drug or placebo were administered to patients in this study.

DETAILED DESCRIPTION:
The inspiratory flow rates achieved by the COPD patients, via the breath actuated devices, are one of the important factors that can influence the efficiency of the drug delivery by the inhalation route. The peak inspiratory flow (PIF) rates achieved by COPD patients through different breath actuated dry power inhalers may differ because of the differences in internal resistance of the different type of devices. The results of inspiratory airflow rate and pressure drop over time, from this study, provided an assessment of the range and variability of inhalation profile characteristics generated by COPD patients within the population selected for this study (e.g. demographics, gender, disease control) through the Breezhaler and the other marketed comparator DPIs.

The inhalation profiles were obtained through an Inhalation Profile Recorder (IPR). The inhalation profile recorder was a data acquisition device which consists of a computer, an interface unit and a pressure transducer. This allowed it to measure the real time dynamic pressure drop at the mouthpiece of the inhaler during an inhalation maneuver. On the graphic user interface, plots of inspiratory pressure drop versus time and flow rate versus time are displayed in real time. The investigator or designated study personnel at site was responsible for typing in the Test Location, selecting the Inhaler Type (Breezhaler, Ellipta, Handihaler), typing in the Patient ID and Patient Age, selecting Male or Female, and recording Patient Comments made during the test session, as necessary.

Each patient were required to generate three (03) inhalational profiles through each of the three (03) study devices: Breezhaler®, Ellipta® and Handihaler®.

ELIGIBILITY:
Inclusion Criteria:

- Current or ex-smokers who have a smoking history of at least 10 pack years (e.g., 10 pack years = 1 pack/day × 10 years, ½ pack/day × 20 years, etc.).

Note: A pack of cigarettes is equal to 20 cigarettes. Occasional smoking of cigars is not relevant to smoking history.

An ex-smoker is defined as a patient who has not smoked for ≥6 months at screening.

* COPD patients with moderate to very severe airflow limitation (spirometric classification: GOLD 2, 3 or 4) at time of screening,

  * Post-bronchodilator FEV1 < 80% of the predicted normal, and
  * Post-bronchodilator FEV1/forced vital capacity (FVC) <0.70. (Post-bronchodilator refers to 1 hour after sequential inhalation of 84 µg ipratropium bromide and 400 µg salbutamol)
* Willing patients assessed as suitable by investigator to reproducibly perform inhalational manoeuvers through study devices as required by the standard protocol
* Willing patients assessed as suitable by investigator to comprehend and follow the instructions for use of the inhalational devices to be tested in the study

Exclusion Criteria:

* Patients with a history of asthma or onset of respiratory symptoms prior to the age of 40 years
* Use of short acting bronchodilating agent (SABA) as rescue (reliever) medication within 6 hours prior to or during inhalational profile assessments for the study [Note: Use of rescue medication should not be restricted if patient feels the need of the rescue/ reliever medication because of the diseased state. Safety and disease management should be priority and the suitability of such a patient for the study or relevance of the (study) assessments done for the study should be reviewed, as appropriate.]
* Patients with any history of premature birth less than 33 weeks gestation or significant level of respiratory care including mechanical ventilation required as neonate affecting the respiratory tract or chronic lung diseases, which in the opinion of the investigator or designated study personnel at site may interfere with the study evaluation or optimal participation in the study.
* Any major chronic illness including but not limited to a diagnosis of non-skin cancer, cystic fibrosis, bronchiectasis, α-1 anti-trypsin deficiency, myelomeningocele, sickle cell anemia, endocrine disease, congenital heart disease, unstable arrhythmia, congestive heart failure, stroke, severe hypertension, insulin-dependent diabetes mellitus, renal failure, liver disorders, immunodeficiency states, significant neurodevelopmental delay or behavioral disorders (excluding mild attention deficit hyperactivity disorder).
* Patients who have had a COPD exacerbation that required treatment with antibiotics or oral corticosteroids or hospitalization in the 6 weeks prior to screening
* Patients who, within 7 days prior to the screening visit (Visit 1) OR prior to Visit 2, increased use of rescue bronchodilators amounting to more than double the average number of puffs used in the preceding week or more than 8 puffs of SABA on any 3 consecutive days or more than 12 puffs of SABA on any 2 consecutive days
* Respiratory tract infections (sinus, middle ear, oropharyngeal, upper or lower respiratory tract infection) within the 4weeks before the visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2016-04-29 (Actual); Study Completion 2016-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma, Study Director — Novartis Pharmaceuticals
Locations (5):
- Argentina (5):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Florida, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As

REFERENCES:
- [Derived] Altman P, Wehbe L, Dederichs J, Guerin T, Ament B, Moronta MC, Pino AV, Goyal P. Comparison of peak inspiratory flow rate via the Breezhaler(R), Ellipta(R) and HandiHaler(R) dry powder inhalers in patients with moderate to very severe COPD: a randomized cross-over trial. BMC Pulm Med. 2018 Jun 14;18(1):100. doi: 10.1186/s12890-018-0662-0. PMID 29898702

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of the 97 screened and randomized patients, 96 patients (99.0%) completed the study.
Pre-assignment Details: No active drug or placebo was administered in this study. The patients were to continue on their respective current maintenance COPD treatment as deemed appropriate by the treating physician. Each patient was required to inhale through all three study devices at the same visit in a randomized cross-over sequence.
Groups:
- Breezhaler/Ellipta/Handihaler; Breezhaler/Handihaler/Ellipta; Ellipta/Breezhaler/Handihaler; Ellipta/Handihaler/Breezhaler; Handihaler/Breezhaler/Ellipta; Handihaler/Ellipta/Breezhaler: Each patient were required to inhale via Breezhaler, Ellipta, and Handihaler in a randomized cross-over sequence. The randomization numbers were generated using 6 sequences: BEH, EHB, HBE, BHE, EBH, HEB (B: Breezhaler, E: Ellipta, H: Handihaler).
Period: Overall Study
Arm/Group | Breezhaler/Ellipta/Handihaler | Breezhaler/Handihaler/Ellipta | Ellipta/Breezhaler/Handihaler | Ellipta/Handihaler/Breezhaler | Handihaler/Breezhaler/Ellipta | Handihaler/Ellipta/Breezhaler
Started | 14 | 16 | 16 | 16 | 18 | 17
Completed | 14 | 15 | 16 | 16 | 18 | 17
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Administrative problems | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Breezhaler/Ellipta/Handihaler
Number analyzed (Participants) | 97
Age, Customized [Number; unit: Years]
  40 - 64 years | 27
  65 - 74 years | 46
  ≥75 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 72

OUTCOME MEASURES:

1. Primary Outcome: Peak Inspiratory Flows Rates Summary by Inhalation Devices - PPS
Description: The peak inspiratory flows (PIF) rates obtained from the inhalation flow profiles generated by the COPD patients through the three dry powder inhalation (DPI) devices(Breezhaler®, Ellipta® and Handihaler®) were measured and compared (without drug or placebo administration). Each patient were required to generate inhalation flow profiles through all three DPI devices in a randomized cross-over sequence. The inspiratory measurements were taken in each of these devices in the same visit.
Time Frame: Visit 2 (Day 1)
Population: Per-protocol set (PPS): This PPS population consisted of all randomized patients, who completed inhalation flow maneuvers through all three inhaler devices.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Breezhaler® | Ellipta® | Handihaler®
Number analyzed (Participants) | 93 | 88 | 93
L/min | 107.52 (23.335) | 80.73 (18.440) | 53.59 (20.629)
Statistical Analysis 1: Comparison: Breezhaler® vs Ellipta®; Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Final Values) = 26.97, 95% CI 2-sided [23.70 to 30.24]
Statistical Analysis 2: Comparison: Breezhaler® vs Handihaler®; Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Final Values) = 53.93, 95% CI 2-sided [49.15 to 58.72]

2. Primary Outcome: Peak Inspiratory Flows Rates Summary by Inhalation Devices - FAS
Description: The peak inspiratory flows (PIF) rates obtained from the inhalation flow profiles generated by the COPD patients through the three dry powder inhalation (DPI) devices(Breezhaler®, Ellipta® and Handihaler®) were measured and compared (without drug or placebo administration). Each patient were required to generate inhalation flow profiles through all three DPI devices in a randomized cross-over sequence. The inspiratory measurements were taken in each of these devices in the same visit.
  This FAS dataset includes PIF data from additional patients with corrected inhaler internal resistance values.
Time Frame: Visit 2 (Day 1)
Population: Full Analysis Set (FAS): The FAS set consisted of all randomized patients who carried out inhalation maneuver through at least one inhaler.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Breezhaler® | Ellipta® | Handihaler®
Number analyzed (Participants) | 97 | 91 | 97
L/min | 108 (23) | 78 (15) | 49 (9)

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse Events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Description: Adverse events were collected without regard to intervention
Arm/Group | Breezhaler/Ellipta/Handihaler
Serious Adverse Events (participants affected / at risk) | 0/97
Other Adverse Events (participants affected / at risk) | 0/97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.